CLINICAL TRIAL: NCT01665352
Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Parallel Group Study to Evaluate the Safety and Efficacy of TTP054 for 12 Weeks in Subjects With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin
Brief Title: A Study to Evaluate Safety and Efficacy of TTP054 for 12 Weeks in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: vTv Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TTP054-201
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- TTP054 400 mg (Experimental)
  Interventions: Drug: TTP054
- TTP054 200 mg (Experimental)
  Interventions: Drug: TTP054
- TTP054 800 mg (Experimental)
  Interventions: Drug: TTP054
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TTP054 — Administered orally once daily for 12 weeks.
  Arms: TTP054 200 mg; TTP054 400 mg; TTP054 800 mg
Drug: Placebo — Administered orally once daily for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety and effect of TTP054 versus placebo on glucose control in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus
* On a stable (for the last 3 months) regimen of either metformin alone or metformin in combination with one additional acceptable oral antidiabetic (OAD) agent
* HbA1c: Metformin only: 7.0 - 11.0%; Metformin + acceptable OAD agent: 6.5 - 9.5%

Exclusion Criteria:

* History or evidence of significant diabetic complications
* History of heart attack, stroke or congestive heart failure
* Severe, uncontrolled hypertension
* Frequent hypoglycemia
* Women of child-bearing potential

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c (%) as compared to placebo | Day 1 to Day 84

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose (mg/dL) | Day 1, Day 14, Day 28, Day 56 and Day 84
Subject achievement of HbA1c <7% | Day 84
Change from baseline in body weight | Day 1, Day 14, Day 28, Day 56 and Day 84
Subject achievement of body weight loss ≥ 2% | Day 1 and Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Gustavson, Ph.D., Study Director — TransTech Pharma, Inc.
Locations (19):
- United States (19):
  - Site 18, Chula Vista, California
  - Site 1, Los Angeles, California
  - Site 13, Denver, Colorado
  - Site 4, Coral Gables, Florida
  - Site 5, Port Orange, Florida
  - Site 3, Honolulu, Hawaii
  - Site 17, Indianapolis, Indiana
  - Site 7, Louisville, Kentucky
  - Site 8, Auburn, Maine
  - Site 9, Las Vegas, Nevada
  - Site 26, Trenton, New Jersey
  - Site 12, Rochester, New York
  - Site 14, Cincinnati, Ohio
  - Site 6, Mt. Pleasant, South Carolina
  - Site 16, Dallas, Texas
  - Site 10, Houston, Texas
  - Site 2, Houston, Texas
  - Site 11, Katy, Texas
  - Site 15, Richmond, Virginia